CLINICAL TRIAL: NCT00265876
Title: A Phase I/II Study of AZD0530 in Combination With Gemcitabine in Patients With Advanced Pancreatic Cancer
Brief Title: AZD0530 and Gemcitabine in Locally Advanced/Metastatic Pancreatic Cancer That Cannot Be Removed By Surgery
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: NCIC Clinical Trials Group (Network)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I173; CAN-NCIC-IND173 (Other: PDQ); ZENECA-CAN-NCIC-IND173 (Other: ASTRAZENECA); CDR0000450844 (Other: PDQ)
Record Dates: First submitted 2005-12-14; First posted 2005-12-15 (Estimated); Last update posted 2023-08-04 (Actual); Status verified 2020-04

CONDITIONS: Pancreatic Cancer
Keywords: adenocarcinoma of the pancreas; stage III pancreatic cancer; recurrent pancreatic cancer; stage IV pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — saracatinib; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AZD0530 + Gemcitabine (Experimental)
  Interventions: Drug: AZD0530; Drug: gemcitabine hydrochloride

INTERVENTIONS:
Drug: AZD0530 — Taken daily every 4 weeks
Drug: gemcitabine hydrochloride — 1000mg/m2 IV weekly

SUMMARY:
RATIONALE: AZD0530 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as gemcitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving AZD0530 together with gemcitabine may kill more tumor cells.

PURPOSE: This phase I/II trial is studying the side effects and best dose of AZD0530 when given together with gemcitabine and to see how well they work in treating patients with locally advanced or metastatic pancreatic cancer that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Phase I

* Determine the maximum tolerated dose of AZD0530 when given in combination with gemcitabine in patients with unresectable, locally advanced or metastatic pancreatic cancer.
* Determine the safety and tolerability of this regimen in these patients.
* Determine toxicity profile and dose-limiting toxicity of this regimen in these patients.
* Determine pharmacokinetic profile of this regimen in these patients.
* Correlate the toxicity profile with the pharmacokinetics of this regimen in these patients.

Phase II

* Determine the objective response rate (partial and complete response) and prolonged stable disease rate in patients treated with this regimen.
* Determine the median survival, 1-year survival, response or stable disease duration, time to disease progression, clinical benefit response, and progression-free survival of patients treated with this regimen.
* Determine the toxicity of this regimen in these patients.
* Correlate changes in serum CTX levels (post-treatment vs baseline) with response and other clinical outcomes in patients treated with this regimen.

OUTLINE: This is a phase I, open-label, multicenter, dose-escalation study of AZD0530 followed by a phase II study.

* Phase I: Patients receive oral AZD0530 once daily on days 1-28 and gemcitabine IV over 30 minutes on days 1, 8, and 15. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients receive 2 additional courses after achieving complete response or stable partial response. Patients with ongoing stable disease receive up to 6 courses. Patients who discontinue gemcitabine due to unacceptable toxicity or who complete 6 courses of therapy may continue to receive AZD0530 alone in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of AZD0530 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. At least 6 patients are treated at the MTD.

* Phase II: Patients receive AZD0530 at the MTD determined in phase I and gemcitabine as in phase I.

After completion of study treatment, patients are followed periodically.

PROJECTED ACCRUAL: A total of 60 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed pancreatic adenocarcinoma

  * Unresectable disease
  * Locally advanced or metastatic disease
* Clinically or radiologically documented disease

  * Measurable or evaluable disease (phase I)
  * Measurable disease, defined as ≥ 1 unidimensionally measurable lesion ≥ 20 mm by conventional techniques OR ≥ 10 mm by spiral CT scan (phase II)

    * Measurable lesion must be outside of previously irradiated field if it is the sole site of disease unless there is documented disease progression
* No known brain metastases

PATIENT CHARACTERISTICS:

Performance status

* ECOG 0-2

Life expectancy

* More than 12 weeks

Hematopoietic

* Platelet count ≥ 100,000/mm^3
* Absolute granulocyte count ≥ 1,500/mm^3

Hepatic

* Bilirubin normal
* AST and ALT ≤ 2 times upper limit of normal (ULN) (5 times ULN if clearly attributable to liver metastasis)

Renal

* Creatinine normal

Cardiovascular

* No active cardiomyopathy
* No congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* No uncontrolled hypertension
* No myocardial infarction within the past 12 months

Pulmonary

* No pulmonary disease requiring oxygen supplementation

Gastrointestinal

* Must not require IV hyperalimentation
* No uncontrolled inflammatory gastrointestinal (GI) disease (e.g., Crohn's disease or ulcerative colitis)
* No active peptic ulcer disease
* No postsurgical malabsorption characterized by uncontrolled diarrhea that results in weight loss and vitamin deficiency
* No other GI tract disease resulting in an inability to take oral medications
* Must be able to take oral medication without crushing, dissolving, or chewing tablets
* Pancreatic enzyme supplementation allowed provided the above conditions are met

Immunologic

* No immune deficiency
* No active, uncontrolled, or serious infection
* No know hypersensitivity to study drugs or their components
* No known HIV positivity

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No history of psychiatric illness (e.g., uncontrolled psychotic disorders) or neurologic disorder that would preclude study compliance
* No other serious medical condition or illness that would preclude study participation
* No other malignancy within the past 5 years except curatively treated nonmelanomatous skin cancer or carcinoma in situ of the cervix or bladder

PRIOR CONCURRENT THERAPY:

Chemotherapy

* No prior chemotherapy except fluorouracil (with or without leucovorin calcium) or gemcitabine given concurrently with radiotherapy as a radiosensitizer

  * At least 4 weeks since prior fluorouracil or gemcitabine

Endocrine therapy

* Concurrent systemic hormonal therapy for symptom control (e.g., appetite stimulation, pain, or nausea) allowed

Radiotherapy

* See Disease Characteristics
* See Chemotherapy
* At least 4 weeks since prior radiotherapy for local disease and recovered

Surgery

* At least 3 weeks since prior major surgery

Other

* At least 2 weeks since prior anticancer therapy or investigational agents
* The following drugs must not be used for 1-2 weeks before, during, and for 1-2 weeks after completion of study treatment:

  * Ketoconazole
  * Itraconazole
  * Ritonavir
  * Mibefradil
  * Clarithromycin
  * Saquinavir mesylate
  * Indinavir sulfate
  * Erythromycin
  * Nefazodone hydrochloride
  * Fluconazole
  * Diltiazem hydrochloride
  * Alfentanil hydrochloride
  * Carbamazepine
  * Cyclosporine
  * Tacrolimus
  * Lovastatin
  * Simvastatin
  * Any other drug known to be a potent inhibitor of cytochrome 3A4
* No other concurrent anticancer therapy or investigational agents

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2006-04-26 (Actual); Primary Completion 2009-01-08 (Actual); Study Completion 2012-01-06 (Actual)

PRIMARY OUTCOMES:
Response (complete [CR] and partial response [PR] or stable disease [SD]) at 8 weeks | 4 years
  Response is assessed every other cycle and will be reported on at final analysis

SECONDARY OUTCOMES:
Toxicity | 4 years
  Toxicity is assessed from the time of first treatment and final results will be reported at final analysis

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm J. Moore, MD, Study Chair — Princess Margaret Hospital, Canada; Sharlene Gill, MD, Study Chair — British Columbia Cancer Agency
Locations (4):
- Canada (4):
  - BCCA - Vancouver Cancer Centre, Vancouver, British Columbia
  - Ottawa Health Research Institute - General Division, Ottawa, Ontario
  - Algoma District Cancer Program, Sault Ste. Marie, Ontario
  - Univ. Health Network-Princess Margaret Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Renouf DJ, Moore MJ, Hedley D, Gill S, Jonker D, Chen E, Walde D, Goel R, Southwood B, Gauthier I, Walsh W, McIntosh L, Seymour L. A phase I/II study of the Src inhibitor saracatinib (AZD0530) in combination with gemcitabine in advanced pancreatic cancer. Invest New Drugs. 2012 Apr;30(2):779-86. doi: 10.1007/s10637-010-9611-3. Epub 2010 Dec 18. PMID 21170669